CLINICAL TRIAL: NCT00730184
Title: Does Potassium Bicarbonate Improve the Effect of Dietary Protein on Bone and Muscle?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Bess Dawson-Hughes, MD, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2510; 7937
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Osteoporosis; Sarcopenia
Keywords: acid-base; potassium; acidosis; osteoporosis; sarcopenia; calcium absorption; dietary protein
MeSH Terms: conditions — Osteoporosis; Sarcopenia; Acidosis | interventions — potassium bicarbonate; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Participants receive potassium bicarbonate in dosage of 90 mmol/d. This compound has no other name.
  Interventions: Dietary Supplement: potassium bicarbonate
- 2 (Placebo Comparator): Participants receive placebo as microcrystalline cellulose. This compound has no other name.
  Interventions: Dietary Supplement: Placebo (microcrystalline cellulose)

INTERVENTIONS:
Dietary Supplement: potassium bicarbonate — 90 mmol/d given as 4 tablets after each meal, with a full glass of water
  Arms: 1
Dietary Supplement: Placebo (microcrystalline cellulose) — Given as 4 tablets after each meal, with a full glass of water
  Arms: 2

SUMMARY:
The purpose of this study is to examine whether adding the basic salt potassium bicarbonate to the diet will have a positive effect on how dietary protein affects your bone and muscle.

DETAILED DESCRIPTION:
The balance between the amount of protein in the diet (anabolic component) and the net acid load of the diet (catabolic component) in part determines whether the diet as a whole has a net anabolic or catabolic effect on bone and muscle. This study will investigate whether the addition of an alkaline salt of potassium, potassium bicarbonate, will allow dietary protein to have a more favorable net impact on intermediary indices of bone and muscle conservation than is observed with protein in the usual acidic environment.

Men and postmenopausal women, age 50 and older, will be enrolled in this 42-day study in order to have 20 completers. Subjects may continue in the study for up to an additional two weeks should this be necessary for reasons related to intercurrent illness (unrelated to the research) or scheduling circumstances. Over the first 15 days, subjects will be placed on gradually increasing doses, up to a maximum of 90 mmol/d of potassium bicarbonate or placebo. They will remain on this dose for the rest of the study. Subjects will then have two 10-day metabolic diet cycles each, in random order, as follows:

Group 1 - low protein diet (0.5 g/kg/d) then high protein diet (1.5 g/kg/d) Group 2 - high protein diet (1.5 g/kg/d) then low protein diet (0.5 g/kg/d)

There will be a 5-day period between the two metabolic diets in which subjects consume their usual diets but continue to take the study pills.

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted in subjects with body mass index < 38 kg/m2.
* Women must be at least 6 months since last menses.
* Subjects must be willing to maintain their usual exercise level and agree not to attempt to gain or lose weight or change their diets substantially during the study.
* Subjects will not be allowed to take their own calcium or vitamin D supplements from one week before their screening visit through the end of the study.
* They must also agree not to ingest bicarbonate- or potassium-rich products such as selected antacids and salt substitutes during the study.
* They must also agree not to consume alcohol during the study.

Exclusion Criteria:

Medications

* Oral glucocorticoid use for > 10 days in the last 3 months
* Estrogen, raloxifene, or calcitonin use in the last 6 months, bisphosphonate or teriparatide use in the last 2 years
* Current use of diuretics
* Regular use of NSAIDS (> 3 times per wk) or anabolic drugs (steroids or other). Note that subjects may use acetominophen for joint or other discomforts during the study.

Conditions/Diseases

* Renal disease including kidney stones in the past 5 years or creatinine clearance < 50 ml/min/1.73 X m2 of body surface area
* Cirrhosis
* GERD requiring treatment with alkali-containing antacids (use of Lowsium okay)
* Hyperparathyroidism
* Untreated thyroid disease
* Significant immune disorder such as rheumatoid arthritis, SLE
* Current unstable heart disease
* Active malignancy or cancer therapy in the last year
* 24-hr urine calcium > 300 mg/d after 1 wk off of calcium supplements
* Subjects with arrythmias (surgically treated arrythmias acceptable), or myocardial infarction in last 12 months
* Total hip T score of < -3.0
* Abnormal serum calcium; alkaline phosphatase >10% above the upper end of the reference range
* Adrenal insufficiency, primary aldosteronism, Bartter's syndrome
* Diabetes mellitus (fasting blood sugar > 130)
* Alcohol use exceeding 2 drinks/day
* Peptic ulcers or esophageal stricture
* Screening serum 25(OH)D levels below 16 ng/ml
* Vegetarians
* Other abnormalities in screening labs, at discretion of the study physician (principal investigator)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To determine the impact of administration of an alkalinizing salt on urinary nitrogen excretion in older men and women. | before and after low and high protein diet cycles
To determine the impact of administration of an alkalinizing salt on urinary calcium excretion in the same population. | before and after low and high protein diet cycle

SECONDARY OUTCOMES:
To determine whether the administration of an alkalinizing salt of potassium alters the effect of protein on biochemical markers of bone turnover in the same population. | before and after low and high protein diet cycles
To determine whether the administration of an alkalinizing salt of potassium alters the effect of protein on calcium absorption in the same population. | before and after low and high protein diet cycles
To determine whether the administration of an alkalinizing salt of potassium alters the effect of protein on serum IGF-1 in the same population. | before and after low and high protein diet cycles

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, MD, Principal Investigator — Tufts University; Lisa Ceglia, MD, Study Director — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ceglia L, Abrams SA, Harris SS, Rasmussen HM, Dallal GE, Dawson-Hughes B. A simple single serum method to measure fractional calcium absorption using dual stable isotopes. Exp Clin Endocrinol Diabetes. 2010 Oct;118(9):653-6. doi: 10.1055/s-0029-1234088. Epub 2009 Oct 23. PMID 19856249